CLINICAL TRIAL: NCT02320123
Title: End-of-Life Care for African Americans: Intervention Design and Implementation
Brief Title: End-of-Life Care for African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ramona L. Rhodes, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STU 032013-051
Record Dates: First submitted 2014-12-15; First posted 2014-12-19 (Estimated); Results first posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Colonic Neoplasms; Breast Neoplasms; Lung Neoplasms
Keywords: Terminal Care; Decision Making; Communication
MeSH Terms: conditions — Colonic Neoplasms; Breast Neoplasms; Lung Neoplasms; Communication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The research staff conducting assessments for all participants was masked to patients receiving the intervention as well as those assigned to the control group.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients - intervention (Experimental): For the intervention arm of the study, patients will be invited to view the educational DVD explaining end-of-life care options and meet with a lay health advisor for discussion.
  Interventions: Behavioral: Educational DVD
- Patients - Control (No Intervention): Patients will receive usual care (nor view the DVD or meet with the lay health advisor).

INTERVENTIONS:
Behavioral: Educational DVD — African American patients and their primary non-professional caregivers will watch a DVD created to introduce end-of-life care planning to African Americans receiving palliative care.
  Arms: Patients - intervention

SUMMARY:
Racial differences in health care are documented across the health care continuum and persist in aging and end-of-life (EOL) care. African Americans (AA) and other underrepresented minorities often choose more aggressive therapies at the end of life and are less likely to utilize hospice care in the terminal stages of their illness. Potential reasons for these disparities include: lack of knowledge of and misperceptions about palliative and hospice care, spiritual beliefs, and mistrust in the health care system, among others. Despite the literature on disparities in end-of-life (EOL) care and reasons for underuse and the presence of national EOL care guidelines, attempts to address this problem have been limited and often not rigorously evaluated. The majority of interventions to promote EOL care were done in majority populations and focused predominantly on trying to change physician awareness of patient's pain, symptoms, and values or to change physician communication behavior. While these early studies made tremendous contributions to the study of EOL care and the needs of the terminally ill, the interventions associated with these studies did not reach their desired effectiveness. The investigators propose a different strategy that would focus specifically on previously identified barriers to utilization of advance directives, palliative care, and hospice care among African Americans - including physicians' difficulty and discomfort with prognostication, AA patients' knowledge, attitudes and beliefs towards hospice and palliative care, conflict between patients' spiritual beliefs and the general hospice and palliative medicine philosophy of care, and medical mistrust. The goal of this project is to improve methods of prognostication for physicians and increase awareness of EOL care options for AAs. To overcome the dual challenges of physicians' reluctance to discuss EOL care and patients' discomfort in engaging in such conversations, the investigators will use the electronic medical record (EMR) to automatically identify AA patients with life-limiting illness who are eligible for counseling about EOL care options. To change knowledge and attitudes toward EOL care options among AA patients, the investigators will design a culturally sensitive intervention that will combine multimedia materials and a culturally concordant lay health advisor who will deliver tailored education and counseling.

DETAILED DESCRIPTION:
Aim 1:

A. We will conduct semi-structured interviews with patient/caregiver pairs and focus groups with providers that will test the communication strategies of available audiovisual materials and materials that we will develop for the intervention. The audiovisual segments will be taken from an available EOL care educational digital versatile disc (DVD). We aim to interview 12 patients and their caregivers, or more until thematic saturation is reached. We will obtain informed consent, and all interviews will be audiotaped and transcribed. Interviews will be conducted separately, and will last 30 to 45 minutes.

B. Two focus groups will be conducted with palliative care providers to identify communication strategies they use with AAs. One will be conducted with providers from Parkland Hospital. The other will be conducted with providers from University Hospitals, the Dallas VA, and Baylor University Medical Center in Dallas. Informed consent will be obtained. All sessions will be audiotaped and transcribed. The focus groups will last 45 to 60 minutes.

C. We will create additional DVD segments that will address previously identified barriers to EOL care for AAs, including: 1) spiritual/religious conflict, and 2) medical mistrust. We will obtain feedback on the newly developed segments from 10 new patient/caregiver dyads (semi-structured interviews) and 6 to 8 AA religious leaders (focus group) recruited from local churches. Informed consent will be obtained prior to conducting the interviews and focus groups. All will last 30 to 60 minutes.

D. A lay health advisor (LHA) will be recruited from the community to provide counsel about EOL care to patients who will receive the intervention. The LHA and the PI of the project will undergo training in how to provide culturally sensitive EOL care for AAs via the APPEAL (A Progressive Palliative Care Educational Curriculum for the Care of AAs at Life's End) Curriculum created at Duke University. After training, the LHA will participate in in-service work with the Parkland Palliative Care Team and the PI.

Aim 2:

We will use an e-EOL algorithm to identify AA patients hospitalized at Parkland who have advanced breast, lung, and colorectal cancer to identify potentially eligible candidates for the intervention utilizing EMR data from Parkland Hospital (See Aim 1 eligibility criteria). Once eligibility is confirmed the LHA will introduce the study to the patient and obtain informed consent. Each patient will be asked to identify a primary caregiver that will be able to participate in the intervention. The LHA will contact the patients' primary caregivers to confirm participation in the study and arrange a time to meet with both the patient and caregiver to conduct the intervention. We anticipate that 24 patient-caregiver pairs will receive the intervention (8 for each type of cancer).

The LHA will meet with eligible patients and caregivers and assist them in watching the developed DVD segments. Afterward, the LHA will answer questions and provide additional information. They will tailor the discussion to the patient's values, preferences, concerns, and clinical circumstances.

The primary process outcome tested will be the feasibility and acceptability of the intervention. Feasibility success will be measured by the number and rates of patients/caregivers who complete the intervention and follow-up interviews. The primary decision-making outcome is change in intent to discuss EOL care options based on the Transtheoretical Stages of Change Model (i.e., pre-contemplation, contemplation, preparation, and action). Secondary outcomes measured will include: knowledge of prognosis and EOL care options, decisional conflict, quality of life, and health care utilization. Other patient and treatment variables will also be collected, per the study protocol.

ELIGIBILITY:
Inclusion Criteria:

Aim 1 patients must:

1. receive their care at Parkland and be diagnosed with advanced cancer (breast, lung, or colon);
2. self-identify as AA;
3. be proficient in English;
4. be competent to give informed consent; and
5. have no evidence of cognitive impairment (Mini-Cog score of ≥3 or 1-2 with normal clock draw).

Aim 2 Patients must:

1. be hospitalized at Parkland
2. be diagnosed with advanced cancer (breast, lung, or colon)
3. self-identify as AA;
4. be proficient in English;
5. be competent to give informed consent;
6. have no evidence of cognitive impairment (Mini-Cog score of ≥3 or 1-2 with normal clock draw); and
7. have never received palliative or hospice care.

All Caregivers (Aim 1 and 2) must be:

1. identified by the selected patients as their primary caregiver;
2. be 21 years of age or older;
3. proficient in English; and
4. competent to give informed consent.

For the expert provider focus group, participants must be a health care provider (physician, nurse practitioner, chaplain, social worker, nurse) who works within hospice and palliative medicine.

(Note: patients who enter palliative care or hospice during follow-up interviews will be allowed to remain in the study)

Exclusion Criteria:

For patients:

1. identify with a race other than African American or
2. have a diagnosis other than advanced breast, lung, or colorectal cancer.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-05-23; Primary Completion 2017-08-10 (Actual); Study Completion 2017-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ethan Halm, MD, Study Director — Chair, Department of General Internal Medicine
Locations (1):
- Parkland Hospital, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients - Intervention: For the intervention arm of the study, patients will be invited to view the DVD explaining end-of-life care options and meet with a lay health advisor for discussion.
  Educational DVD: African American patients and their primary non-professional caregivers will watch a DVD created to introduce end-of-life care planning to African Americans receiving palliative care.
- Patients - Control: For the control arm of the study, patients will receive usual care (not view the DVD or meet with the lay health advisor).
  Usual Care
Period: Overall Study
Arm/Group | Patients - Intervention | Patients - Control
Started | 10 | 12
Completed | 0 | 1
Not Completed | 10 | 11
Not completed — Lost to Follow-up | 4 | 6
Not completed — Death | 6 | 5

BASELINE CHARACTERISTICS:
Population: One patient initially assigned to the control group was deemed ineligible and was removed from the study, leaving 12 patients assigned to the control group for analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients - Intervention | Patients - Control | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 14
  >=65 years | 4 | 4 | 8
Age, Continuous [Mean (Full Range); unit: years] | 60.4 [36 to 78] | 58.6 [36 to 75] | 59.4 [36 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 12 | 22
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 12 | 22
Hospitalized patients with cancer [Count of Participants; unit: Participants] | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Intent to Discuss Advance Directives (Based on the Transtheoretical Stages of Change Model)
Description: The primary decision-making outcome is change in intent to discuss advance directives based on the Transtheoretical Stages of Change Model (i.e., pre-contemplation, contemplation, preparation, action, and maintenance).
Time Frame: Within six months after patient enrolls in study, June 2017.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients - Intervention | Patients - Control
Number analyzed (Participants) | 10 | 12
Participants
  Pre-contemplation | 0 | 1
  Contemplation | 1 | 3
  Preparation | 2 | 4
  Action | 0 | 0
  Maintenance | 4 | 0
  Participant doesn't know | 3 | 4

2. Primary Outcome: Intent to Discuss Medical Power of Attorney (Based on the Transtheoretical Stages of Change Model)
Description: The primary decision-making outcome is change in intent to discuss medical power of attorney based on the Transtheoretical Stages of Change Model (i.e., pre-contemplation, contemplation, preparation, action, and maintenance).
Time Frame: Within six months after patient enrolls in study, June 2017.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients - Intervention | Patients - Control
Number analyzed (Participants) | 10 | 12
Participants
  Pre-contemplation | 0 | 3
  Contemplation | 3 | 1
  Preparation | 2 | 5
  Action | 0 | 1
  Maintenance | 2 | 0
  Participant doesn't know | 3 | 2

3. Primary Outcome: Intent to Discuss Palliative Care (Based on the Transtheoretical Stages of Change Model)
Description: The primary decision-making outcome is change in intent to discuss palliative care based on the Transtheoretical Stages of Change Model (i.e., pre-contemplation, contemplation, preparation, action, and maintenance).
Time Frame: Within six months after patient enrolls in study, June 2017.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients - Intervention | Patients - Control
Number analyzed (Participants) | 10 | 12
Participants
  Pre-contemplation | 2 | 4
  Contemplation | 2 | 2
  Preparation | 1 | 1
  Action | 2 | 3
  Maintenance | 0 | 0
  Participant doesn't know | 3 | 2

4. Primary Outcome: Intent to Discuss Hospice Care (Based on the Transtheoretical Stages of Change Model)
Description: The primary decision-making outcome is change in intent to discuss hospice care based on the Transtheoretical Stages of Change Model (i.e., pre-contemplation, contemplation, preparation, action, and maintenance).
Time Frame: Within six months after patient enrolls in study, June 2017.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients - Intervention | Patients - Control
Number analyzed (Participants) | 10 | 12
Participants
  Pre-contemplation | 7 | 10
  Contemplation | 1 | 1
  Preparation | 1 | 0
  Action | 0 | 0
  Maintenance | 0 | 0
  Participant doesn't know | 1 | 1

5. Secondary Outcome: Quality of Life at the End of Life
Description: This will be assessed by using the McGill QOL Questionnaire, Part A, which measures overall quality of life in a 48 hour period: "Considering all parts of my life - physical, emotional, social, spiritual, and financial - over the past two (2) days the quality of my life has been: 0-10," with 0=very bad and 10=excellent.
Time Frame: Within six months after patient enrolls in study, June 2017.
Population: All study participants were assessed by using the McGill QOL questionnaire
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Patients - Intervention | Patients - Control
Number analyzed (Participants) | 10 | 12
score on a scale | 6.4 [3.68 to 9.12] | 6.1 [3.67 to 8.50]

6. Secondary Outcome: Health Care Utilization: Emergency Room
Description: Health care utilization will be measured mean number of ER visits for the intervention and control groups.
Time Frame: Within six months after patient enrolls in study, June 2017.
Measure: Mean (95% Confidence Interval); unit: ER Visits
Groups:
- Intervention Group: For the intervention arm of the study, patients will be invited to view the DVD explaining end-of-life care options and meet with a lay health advisor for discussion.
  Educational DVD: African American patients and their primary non-professional caregivers will watch a DVD created to introduce end-of-life care planning to African Americans receiving palliative care.
- Control Group: For the control arm of the study, patients will receive usual care (not view the DVD or meet with the lay health advisor).
  Usual Care
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 10 | 12
ER Visits | 4.5 [0.91 to 8.08] | 2.5 [0.55 to 4.44]

7. Secondary Outcome: Number of Patients Who Died
Description: The principal investigator or research staff will attempt to determine the date and location of death for patients who have died while enrolled in the study by reviewing the patient's electronic health record.
Time Frame: Within six months after patient enrolls in study, June 2017.
Population: Deceased at six months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients - Intervention | Patients - Control
Number analyzed (Participants) | 10 | 12
Participants | 6 | 6

8. Secondary Outcome: Utilization of Advance Care Planning and End-of-life Care
Description: The number of participants who have documentation of advance care planning, palliative care clinic visits, and/or hospice enrollment.
Time Frame: Within six months after patient enrolls in study, June 2017.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients - Intervention | Patients - Control
Number analyzed (Participants) | 10 | 12
Participants
  Documentation of enrollment in hospice | 3 | 3
  Documentation of medical power of attorney | 4 | 4
  Documentation of living will | 1 | 0
  Documentaon of palliative care | 4 | 4
  Deceased | 6 | 6

9. Secondary Outcome: Health Care Utilization: Mean Number of Hospitalizations in Six Months by Group
Description: Health care utilization will be measured mean number of hospitalizations by group, obtained by chart abstraction.
Time Frame: Within six months after patient enrolls in study, June 2017.
Measure: Mean (95% Confidence Interval); unit: Hospitalizations
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 10 | 12
Hospitalizations | 4.2 [1.3 to 7.09] | 2.2 [.71 to 3.62]

ADVERSE EVENTS:
Time Frame: 1 year
Description: The study procedures do not involve any medical procedures or interventions. Procedures are limited to patients answering survey questions, and patients randomized to the intervention arm will view an educational video. Because eligible patients must have a diagnosis of advanced cancer, it's possible some patients my die prior to completing study surveys ("all-cause mortality"). In addition, patients may experience psychological distress answering survey questions ("other").
Arm/Group | Patients - Intervention | Patients - Control
All-Cause Mortality (participants affected / at risk) | 6/10 | 6/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 0/10 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2017-01-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT02320123/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/23/NCT02320123/Prot_SAP_001.pdf